CLINICAL TRIAL: NCT05965882
Title: A Registry Study of Biomarkers in Ischemic Heart Disease ( BIOMS-IHD )
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Collaborators: Beijing Luhe Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: BIOMS-IHD
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Cardiovascular Diseases
Keywords: Ischemic heart disease
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The registry study aims to discover biomarkers for accurate classification and risk assessment of ischemic heart disease.

DETAILED DESCRIPTION:
The purpose of this study is to discover biomarkers for early identification, diagnosis, molecular classification, and intervention based on the mechanism of ischemic heart disease（IHD）. Using mass spectrometry-based metabolomics and multimodal imaging technology, the study aims to further construct a new system for early risk stratification of IHD based on abnormal metabolites.

ELIGIBILITY:
Inclusion criteria :

* Aged 18 years or older.
* Previous ischemic symptoms/signs or electrocardiographic ischemic changes and.
* >70% stenosis of at least one epicardial coronary artery on angiography or a history of myocardial infarction or coronary revascularization.

Exclusion Criteria:

* Current known inability to follow instructions or comply with follow-up procedures.
* Eligible patients without informed consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Partients with ischemic heart disease accorrding to Inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Number of hospitalizations for acute heart failure (HF) | These data is collected during follow-up visit at 3/6/12/24/36/48 months after discharge
  Unplanned emergency visits or hospitalizations leading to HF deterioration were defined as hospitalizations for HF

SECONDARY OUTCOMES:
Number of major adverse cardiovascular events (MACE) | These data is collected during follow-up visit at 3/6/12/24/36/48 months after discharge
  Major adverse cardiovascular events (MACE) in overall population, defined as composite of all-cause death, Heart Failure hospitalization, recurrent myocardial infarction, stroke or ischemia-driven revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Du, phD, Study Director — The Key Laboratory of Remodeling-Related Cardiovascular Disease, Ministry of Education, Beijing Anzhen Hospital, Capital Medical University, Beijing Institute of Heart,Lung and Blood Vessel Diseases
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China